CLINICAL TRIAL: NCT04627779
Title: The Effect of Sex Difference in Preemptive Analgesic Effects With Flurbiprofen Axetil on Postoperative Pain and Sleep Quality of Patients Under General Anesthesia
Brief Title: Sex Difference in Preemptive Analgesic Effects With Flurbiprofen Axetil on Postoperative Pain and Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bijia Song, principal investigator, Beijing Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sex difference and pain
Record Dates: First submitted 2020-11-04; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Preemptive Analgesia; Sex Difference; Flurbiprofen Axetil; Postoperative Pain; Postoperative Sleep Quality
MeSH Terms: conditions — Pain, Postoperative | interventions — flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male Group (Experimental)
  Interventions: Drug: preemptive analgesia with flurbiprofen axetil
- Female Group (Active Comparator)
  Interventions: Drug: preemptive analgesia with flurbiprofen axetil

INTERVENTIONS:
Drug: preemptive analgesia with flurbiprofen axetil — give flurbiprofen axetil 15 min before surgery

SUMMARY:
In humans and animals, circadian rhythm sleep cycle plays an important role on maintaining and regulating basic physiological homeostasis, such as cognitive function, glucose metabolism, memory consolidation, immune function and growth hormone secretion. The induction of general anesthesia leads to a state of reduced responsiveness, which is often described by anesthesiologists and patients as "sleep". This seems to be a common problem in the case of patients under general anesthesia, besides surgery trauma and general anesthetics may change sleep function and sleep cycle perioperatively, the postoperative complications such as pain, nausea and vomiting etc after general anesthesia may also reduce postoperative sleep quality.Flurbiprofen axetil is a new non-steroidal anti infection analgesic(NSAIDs), which is widely used for analgesia to reduce the dose of opioids and the occurrence of adverse reactions, such as declined sleep quality, respiratory depression, nausea and vomiting . Preemptive analgesia is an analgesic intervention that begins before surgery to prevent the nervous system from becoming sensitive to subsequent stimuli that may aggravate pain. A large number of experimental studies have shown that use flurbiprofen axetil preoperatively is better than use it postoperatively. However, limited information was reported before on the effect of factors such as age, gender, preoperative negative mood such as anxiety and depression, type and length of surgery, which could influence postoperative pain and analgesic consumption and the association between postoperative sleep quality and postoperative pain intensity. At present, there has been less previous evidence for how preemptive analgesic with flurbiprofen axetil affect postoperative sleep quality through its effect on postoperative pain of patients with different sex under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 80 years;
2. American Society of Anaesthesiologists (ASA) physical status I-Ⅲ.

Exclusion Criteria:

1. patients with central nervous system and mental illness;
2. patients with preoperative sleep disorders;
3. patients with a history of sedation, analgesia or antidepressants;
4. patients with sleep apnea or obstructive sleep apnea hypopnea syndrome;
5. patients with chronic gastritis and gastric ulcer
6. patients who are allergic to flurbiprofen axetil.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 24 hours after surgery
  use Visual analogue scale (VAS) score to evaluate postoperative pain,0 was considered painless, and a score of 10 was considered as intense pain
postoperative sleep distribution (Rapid eye movement, unstable sleep and stable sleep) tested by Portable Sleep Monitor | first night before surgery
  use sleep monitor to evaluate postoperative sleep distribution (Rapid eye movement, unstable sleep and stable sleep)
postoperative sleep distribution (Rapid eye movement, unstable sleep and stable sleep) tested by Portable Sleep Monitor | first night after surgery
  use sleep monitor to evaluate postoperative sleep distribution (Rapid eye movement, unstable sleep and stable sleep)
postoperative sleep distribution (Rapid eye movement, unstable sleep and stable sleep) tested by Portable Sleep Monitor | third night after surgery
  use sleep monitor to evaluate postoperative sleep distribution (Rapid eye movement, unstable sleep and stable sleep)

SECONDARY OUTCOMES:
postoperative adverse effects | 24 hours after surgery
  evaluate postoperative adverse effects